CLINICAL TRIAL: NCT00358722
Title: A Long-term, Open-label Continuation Study to Assess the Safety of Magnesium Iron Hydroxycarbonate in Haemodialysis Subjects With Hyperphosphataemia
Brief Title: An Evaluation of the Long-term Safety of Magnesium Iron Hydroxycarbonate
Acronym: ALCON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited number of subjects
Sponsor: Ineos Healthcare Limited (Industry)
Responsible Party: Chief Medical Officer, Ineos Healthcare Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IH 002 (ALCON)
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — iron-magnesium hydroxycarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fermagate (Experimental)
  Interventions: Drug: Fermagate

INTERVENTIONS:
Drug: Fermagate — Film coated tablet 500mg
  Other Names: Alpharen

SUMMARY:
Fermagate is a phosphate binder that absorbs phosphate from food, reducing the amount that the body can absorb.

The purpose of this study it to look at the safety of fermagate over longer periods of time.

DETAILED DESCRIPTION:
High levels of phosphate in the blood are linked with serious effects, due to calcium imbalances (high levels of parathyroid hormone (PTH), bone disease, formation of calcium deposits in the body, and blood-vessel disease).

This study is an open-label, multi-centre, single-group, 24-week study of fermagatebonate. Subjects participating in this study are those who took at least one dose of double-blind study medication in the IH 001 study and either completed study IH 001 or were withdrawn due to reasons other than an adverse event (AE) considered related to study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Taken at least one dose of double-blind medication during study IH 001 and either completed study IH 001 or were withdrawn due to reasons other than an AE considered related to study treatment
2. Male or female subjects on active haemodialysis, aged 18 years or over
3. Willing to abstain from taking any phosphate binder or oral magnesium-, aluminium-, or iron-containing products and preparations, other than the study medication;
4. Willing to avoid any intentional changes in diet such as fasting, dieting or overeating;
5. Willing to maintain their usual type and dose of Vitamin D supplementation.

Exclusion Criteria:

1. Participation in any other clinical trial using an investigational product or device within the previous 4 months;
2. A significant history of alcohol, drug or solvent abuse in the opinion of the investigator;
3. Any disease or condition, physical or psychological, which in the opinion of the investigator would compromise the safety of the subject or increase the likelihood of the subject being withdrawn;
4. Clinically significant laboratory findings (for this subject population) in the opinion of the investigator.
5. Any malignancy with the exception of basal cell carcinoma;
6. A history of a motility disorder of the intestines, including, but not limited to, gastroparesis, ileus, pseudo-obstruction, megacolon, or mechanical obstruction;
7. A significant illness in the 4 weeks before screening;
8. Taking medication for seizures;
9. A history of haemochromatosis;
10. A history of serum ferritin concentration of ≥ 1000 ng/mL (excluding transient, treatment-induced ferritin elevation);
11. A history of dysphagia or swallowing disorders;
12. Female subjects who are lactating or pregnant. Women of childbearing potential (pre-menopausal and not surgically sterilised) unless they abstain from sexual intercourse or are using a reliable contraceptive method, that is, barrier methods, hormones or intrauterine device;
13. Current haemoglobin concentration of < 10.00 g/dL;
14. Allergy to the IMP or its constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Assessment of AEs and other safety parameters | 88 weeks

SECONDARY OUTCOMES:
Assessment of serum phosphate concentrations | 88 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon Roe, MB ChB, Principal Investigator — Nottingham City Hospital
Locations (15):
- United States (4):
  - 1614 West 42nd Street, Pine Bluff, Arkansas
  - US Renal Care, Stuttgart, Arkansas
  - Davita Dialysis Center, Charlotte, North Carolina
  - Southeast Renal Associates, Charlotte, North Carolina
- United Kingdom (11):
  - Renal Unit, Birmingham Heartlands Hospital, Birmingham
  - St Lukes Hospital, Little Horton Lane, Bradford
  - Richard Bright Renal Unit, Southmead Hospital, Bristol
  - Addenbrookes Dialysis Centre, Addenbrookes Hospital, Cambridge
  - Renal Unit, Leicester General Hospital, Leicester
  - Dialysis Unit, Broad Green Hospital, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - General Medicine and Nephrology, Norfolk and Norwich University Hospital, Norwich
  - Nottingham Renal and Transplant Unit, Nottingham City Hospital, Nottingham
  - Sheffield Kidney Unit, Northern General Hospital, Sheffield
  - Dept. of Nephrology, Morriston Hospital, Swansea